CLINICAL TRIAL: NCT00001178
Title: Regional Cerebral Utilization of Glucose in Patients With a Diagnosis of Frontal Lobe Dementia, Atypical Parkinsonian Disorder, and Other Basal Ganglia Disorders
Brief Title: Brain Study of Patients With Frontal Lobe Dementia and Parkinsonian Disorders
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 810010; 81-N-0010
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-12-17

CONDITIONS: Alzheimer's Disease; Dementia; Down's Syndrome
Keywords: Alzheimer's Disease; Cerebral Metabolism; Cerebrospinal Fluid; Dementia of the Alzheimer Type; 18-F-Fluoro-2-Deoxy-D-Glucose (FDG); Magnetic Resonance Imaging; Positron Emission Tomography; X-Ray Computed Tomography (CT); Senile Dementia; Down Syndrome; Trisomy 21
MeSH Terms: conditions — Alzheimer Disease; Dementia; Down Syndrome

SUMMARY:
The Cognitive Neuroscience Section of the National Institute of Neurological Disorders and Stroke proposes to continue its cross-sectional and longitudinal studies of cerebral metabolism in frontal lobe dementias and atypical basal ganglia disorders. These studies include repeated assessments of neuropsychological and brain anatomical and metabolic function in subjects with these important and possibly related brain disorders.

DETAILED DESCRIPTION:
Objective

To continue the cross-sectional and longitudinal studies performed by the Cognitive Neuroscience Section of NINDS on the neuroanatomy, cerebral metabolism, neuropsychology, and genetics of frontotemporal dementia, corticobasal syndrome, and related brain disorders.

Study population

Frontal lobe dementias and atypical basal ganglia disorders including frontotemporal dementia, corticobasal syndrome, and related brain disorders.

Design

A cross-sectional assessment of neuropsychological, brain anatomical and metabolic function, and genetic measures in subjects with these disorders.

Outcome measures

MRI, FDG-PET, neuropsychological and clinical tests, genetics, and neuropathology.

ELIGIBILITY:
* Subjects will be recruited from the NIH referral center, neurological and psychiatric clinics, from self or family referral in response to advertisements or from private physicians. Healthy volunteers will include subjects who are considered at-risk for the development of FTD or CBS and subjects who serve as normal controls matched for key characteristics with the patients.

INCLUSION CRITERIA FOR PATIENTS:

* Diagnosis of possible / probable FTD or CBS
* Caregiver willing and able to accept the responsibilities involved in the study

EXCLUSION CRITERIA:

* Pregnant women. Women of childbearing potential will be screened by history for the possibility of pregnancy and undergo a urine pregnancy test. These women will be excluded from the imaging portions of the protocol.
* Behavioral symptoms that would preclude the gathering of data for the study
* Other medical or social condition that would preclude participation in the opinion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 1981-01-19; Study Completion 2012-12-17

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schwartz M, Creasey H, Grady CL, DeLeo JM, Frederickson HA, Cutler NR, Rapoport SI. Computed tomographic analysis of brain morphometrics in 30 healthy men, aged 21 to 81 years. Ann Neurol. 1985 Feb;17(2):146-57. doi: 10.1002/ana.410170208. PMID 3872096
- [Background] Schlageter NL, Horwitz B, Creasey H, Carson R, Duara R, Berg GW, Rapoport SI. Relation of measured brain glucose utilisation and cerebral atrophy in man. J Neurol Neurosurg Psychiatry. 1987 Jun;50(6):779-85. doi: 10.1136/jnnp.50.6.779. PMID 3497229
- [Background] Duara R, Grady C, Haxby J, Ingvar D, Sokoloff L, Margolin RA, Manning RG, Cutler NR, Rapoport SI. Human brain glucose utilization and cognitive function in relation to age. Ann Neurol. 1984 Dec;16(6):703-13. doi: 10.1002/ana.410160613. PMID 6335379